CLINICAL TRIAL: NCT05129358
Title: Testing of an Electronic Patch During Dehydration in Healthy Volunteers
Brief Title: Testing of an Electronic Patch During Mild Dehydration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mode Sensors AS (Industry)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CTR041 REO
Record Dates: First submitted 2021-10-29; First posted 2021-11-22 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Dehydration
Keywords: Dehydration; Rehydration
MeSH Terms: conditions — Dehydration | interventions — Fluid Therapy

STUDY DESIGN:
Intervention Model Description: Open-labeled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hydration sensor (Experimental): The subjects use the wearable hydration sensor for ten days and undergo a dehydration/rehydration intervention on day 2 or 3.
  Interventions: Drug: Dehydration; Dietary Supplement: Rehydration

INTERVENTIONS:
Drug: Dehydration — The subject is brought to mild dehydration (loss of approximately 1.5% of body weight) through intravenous injection of up to 40 ug Furosemide. The subject shall not ingest any fluid for the next 120 minutes.
  Other Names: Dehydration from Furosemide
Dietary Supplement: Rehydration — The subject is rehydrated by oral intake of 1.5 liters Resorb Sport (Nestlé). The subject is monitored for 60 minutes following intake.
  Other Names: Rehydration by Resorb Sport

SUMMARY:
The purpose of this study is to investigate the ability of a wearable bioimpedance sensor to detect mild dehydration in healthy volunteers following the administration of Furosemide. In addition, the study will investigate changes in bioimpedance related to normal variation in tissue hydration (circadian changes, skin thickness, posture, and moderate activity). The study will also provide information on the durability of the sensor.

DETAILED DESCRIPTION:
The subjects will use the patches for ten days. During the ten-day period, subjects are exposed to an intervention on day 2 or 3 while being monitored by health personnel:

* Subjects are given a diuretic (Furosemide) and monitored for two hours without any intake.
* The intervention is followed by intake of a rehydration solution (up to 1500 ml), containing glucose and electrolytes (Resorb Sport, Nestle S.A.).

ELIGIBILITY:
Inclusion Criteria:

* BMI: 18-30
* Age: 18-60
* Willing to refrain from exercise for the duration of the study
* Willing to refrain from bathing, swimming and other physical activity causing considerable sweating/movement (e.g. cycling, mountain hiking, climbing)

Exclusion Criteria:

* Hypersensitivity to diuretics
* Diarrhea
* Hypotension or orthostatic hypotension
* Urinary retention
* Pregnancy or breast feeding
* Allergy to medical adhesive or gel
* Any planned medical examination during the intervention period
* Pacemaker
* Use of medication with a significant impact on the body's fluid balance, such as diuretic

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2023-11-03 (Actual)

PRIMARY OUTCOMES:
Change in impedance following mild dehydration | 2 hours
  Relative change in extracellular resistance measured by the investigational device following administration of Furosemide compared to control days

SECONDARY OUTCOMES:
Change in impedance following rehydration | 1 hour
  Relative change in extracellular resistance measured by the investigational device following ingestion of 1500 ml Resorb (Nestlé)

CONTACTS AND LOCATIONS:
Overall Officials: Sigve N Aas, PhD, Study Director — Mode Sensors AS
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
No sharing planned. Application to ethical board does not include permission to share.

REFERENCES:
- [Derived] Noddeland H, Bremnes F, Thorud A, Rolid K, Kvaerness J, Jaatun EA, Aas SN. A novel wearable bioimpedance sensor for continuous monitoring of fluid balance: a study on isotonic hypovolemia in healthy adults. J Clin Monit Comput. 2025 Apr;39(2):379-391. doi: 10.1007/s10877-024-01245-z. Epub 2024 Dec 4. PMID 39630397